CLINICAL TRIAL: NCT06179810
Title: Effect of Baduanjin Exercise on Quality of Life in Patients With Metabolic Syndrome
Brief Title: Effect of Baduanjin Exercise on Metabolic Syndrome Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed eldeeb, EFFECT OF BADUANJIN EXERCISE ON QUALITY OF LIFE IN PATIENTS WITH METABOLIC SYNDROME, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P. T. REC/012/004558
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: Pre/posttest randomized control trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baduanjin exercise in addition to medical treatment (Experimental): 30 patients with metabolic syndrome do baduanjin exercise in addition to traditional medical treatment
  Interventions: Other: Baduanjin exercise
- Traditional medical treatment (Experimental): 30 patients with metabolic syndrome taking traditional medical treatment
  Interventions: Other: Baduanjin exercise

INTERVENTIONS:
Other: Baduanjin exercise — Baduanjin exercise

SUMMARY:
Pre/posttest randomized control trial design.

In this study all patients will be randomly assigned into two groups (30 in each group) :

* Group A will do baduanjin exercise in addition to traditional medical treatment.
* Group B will take traditional medical treatment only.

ELIGIBILITY:
Inclusion Criteria:

* metabolic syndrome patients

Exclusion Criteria:

* patients with Respiratory diseases
* patients with pacemaker patients
* patients with Neurological diseases
* patients with orthopedic diseases

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Fasting glucose level | 3 months
  Pre/post fasting glucose level in blood
Lipids profile | 3 months
  Pre/post HDL & lDL levels in blood

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Mohamed Abdelrahman Eldeeb, Cairo, Qaliop Elbalad, Egypt